CLINICAL TRIAL: NCT04607135
Title: Acoustic Radiation Force Impulse (ARFI) Imaging for Targeted Prostate Biopsy
Brief Title: ARFI Imaging for Targeted Prostate Biopsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Current sample size sufficiently powers the study to evaluate outcome measures
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00106093
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Transrectal Ultrasound; Prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Elasticity Imaging Techniques; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Acoustic radiation force impulse (ARFI) (Experimental): Patients with suspected PCa who are scheduled to undergo an ultrasound fusion-MR prostate biopsy.
  Interventions: Device: Acoustic radiation force impulse (ARFI)
- MR-ultrasound fusion (Active Comparator): Patients with suspected PCa who are scheduled to undergo an ultrasound fusion-MR prostate biopsy.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Acoustic radiation force impulse (ARFI) — Sound waves are sent in a series and are expected to "push on" the prostate and move it a very small amount (the width of a hair). The stiffer the structure (prostate), the less it will move. This motion will be detected by the ultrasound system
  Arms: Acoustic radiation force impulse (ARFI)
Device: Ultrasound — Standard ultrasound imaging session, ultrasound sound waves are sent into the tissue and bounce off of structures to make an image that appears on a screen
  Arms: MR-ultrasound fusion

SUMMARY:
The purpose of this study is to evaluate a new ultrasound technique. This technique may provide additional and improved information about the stiffness and sizes of the internal structures of your prostate in order to improve the guidance for a targeted biopsy. The investigational, custom-designed probe and needle guide will be used to produce images of your prostate and provide guidance for up to 4 additional biopsy samples (cores) prior to a standard magnetic resonance (MR) ultrasound fusion biopsy procedure. Above the time required for the MR ultrasound fusion biopsy, this study will take up to 30 additional minutes of time for collection of the investigational device guided collection of biopsy samples Risks of participation include increased time under anesthesia (to collect additional biopsies) and slight heating of tissue.

ELIGIBILITY:
Inclusion Criteria:

* Men who are scheduled to undergo ultrasound fusion-MR prostate biopsy;
* Men who are willing to participate in the study;
* Subjects must freely sign informed consent to enroll in the study;
* Assessing eligibility: eligibility for the study will be assessed, based upon the above criteria, by the participating urologist at the time of consultation.
* 18 years or older

Exclusion Criteria:

* Men who have had previous treatment for PCa including radiation, cryoablation, chemotherapy, surgery, high intensity focused ultrasound (HIFU), laser therapy or hormone therapy;
* Men who have had previous non-pharmacological invasive or minimally invasive treatment for benign prostatic hypertrophy (BPH) (i.e., TURP, TUMPT, WIT, TUNA, etc);
* standard pharmacological treatment of BPH is allowable
* Men who are mentally impaired and cannot give written consent;
* Men with anomalies of the rectum.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Polascik, MD, Principal Investigator — Duke University; Kathryn Nightingale, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan DY. A 3-D Multiparametric Ultrasound Elasticity Imaging System for Targeted Prostate Biopsy Guidance [dissertation]. Durham (NC): Duke University; 2023.
- [Result] Chan DY, Moavenzadeh SR, Wightman WE, Palmeri ML, Polascik TJ, Nightingale KR. Clinical Feasibility of 3-D Acoustic Radiation Force Impulse (ARFI) Imaging for Targeted Prostate Biopsy Guidance. Ultrason Imaging. 2025 Mar;47(2):79-92. doi: 10.1177/01617346241311901. Epub 2025 Jan 6. PMID 39760302
- [Result] Moavenzadeh SR, Chan DY, Adams ES, Deivasigamani S, Kotamarti S, Palmeri ML, Polascik TJ, Nightingale KR. Evaluation of 3D ARFI imaging of prostate cancer: diagnostic reliability and concordance with MpMRI. Cancer Imaging. 2025 Apr 23;25(1):55. doi: 10.1186/s40644-025-00874-0. PMID 40270056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study took place from October 2021 to March 2023.
Pre-assignment Details: Record and results are representative of Part 2 of the protocol. The results of Part 1 were not intended to be reported with Part 2.
Groups:
- Patients With Suspected PCa Who Are Scheduled to Undergo an Ultrasound Fusion-MR Prostate Biopsy: Acoustic radiation force impulse (ARFI): Sound waves are sent in a series and are expected to "push on" the prostate and move it a very small amount (the width of a hair). The stiffer the structure (prostate), the less it will move. This motion will be detected by the ultrasound system. Regions suspicious for cancer in ARFI images are biopsied under ARFI imaging guidance.
  Ultrasound: Standard ultrasound imaging session, ultrasound sound waves are sent into the tissue and bounce off of structures to make an image that appears on a screen. MR fusion methods are used to provide imaging guidance to target biopsies.
  Systematic sampling: Biopsy specimens are obtained by sampling 12 pre-specified locations in the prostate, with standard ultrasound imaging guidance.
Period: Overall Study
Arm/Group | Patients With Suspected PCa Who Are Scheduled to Undergo an Ultrasound Fusion-MR Prostate Biopsy
Started | 34
Acoustic Radiation Force Impulse (ARFI) | 30
MR-ultrasound Fusion | 29
Systematic Sampling | 30
Completed | 29
Not Completed | 5
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Equipment not working | 3

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Suspected PCa Who Are Scheduled to Undergo an Ultrasound Fusion-MR Prostate Biopsy
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Whom the Biopsy Approach Detected the Presence of Prostate Cancer (PCa) of Any Grade
Time Frame: Up to 30 minutes
Population: Participants who were imaged with that biopsy approach and in whom cancer of any grade was detected by any biopsy approach. All but one participant underwent all three types of biopsy. One subject did not undergo MR-ultrasound fusion biopsy, but did complete the other two procedures.
Measure: Count of Participants; unit: Participants
Groups:
- Acoustic Radiation Force Impulse (ARFI): Patients with suspected PCa who are scheduled to undergo an ultrasound fusion-MR prostate biopsy.
  Acoustic radiation force impulse (ARFI): Sound waves are sent in a series and are expected to "push on" the prostate and move it a very small amount (the width of a hair). The stiffer the structure (prostate), the less it will move. This motion will be detected by the ultrasound system. Regions suspicious for cancer in ARFI images are biopsied under ARFI imaging guidance.
- MR-ultrasound Fusion: Patients with suspected PCa who are scheduled to undergo an ultrasound fusion-MR prostate biopsy.
  Ultrasound: Standard ultrasound imaging session, ultrasound sound waves are sent into the tissue and bounce off of structures to make an image that appears on a screen. MR fusion methods are used to provide imaging guidance to target biopsies.
- Systematic Sampling: Patients with suspected PCa who are scheduled to undergo an ultrasound fusion-MR prostate biopsy.
  Systematic sampling: Biopsy specimens are obtained by sampling 12 pre-specified locations in the prostate, with standard ultrasound imaging guidance.
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 27 | 26 | 27
Participants | 13 | 22 | 23

2. Primary Outcome: Length of Cancerous Tissue
Description: Length of carcinoma per cancer-positive biopsy specimen as reported by the pathology findings, computed from all cancer-positive biopsy specimens from a given biopsy approach for each participant in whom cancer of any grade was detected by any biopsy approach.
Time Frame: Up to 30 minutes
Population: Participants in whom cancer was detected by a given biopsy approach.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 13 | 22 | 23
mm | 9.5 (11.2) | 15.8 (10.3) | 4.9 (3.0)
Statistical Analysis 1: Comparison: Acoustic Radiation Force Impulse (ARFI) vs MR-ultrasound Fusion vs Systematic Sampling; Test type: Other; p = 0.0003, Welch's ANOVA — F-statistic = 11.71
Statistical Analysis 2: Comparison: MR-ultrasound Fusion vs Systematic Sampling; Test type: Other; p = 0.002, Games-Howell post-hoc test — q-statistic = 6.74
Statistical Analysis 3: Comparison: Acoustic Radiation Force Impulse (ARFI) vs MR-ultrasound Fusion; Test type: Other; p = 0.24, Games-Howell post-hoc test — q-statistic = 2.34
Statistical Analysis 4: Comparison: Acoustic Radiation Force Impulse (ARFI) vs Systematic Sampling; Test type: Other; p = 0.35, Games-Howell post-hoc test — q-statistic = 2.04

3. Primary Outcome: Grade Group of Cancerous Tissue
Description: The grading system has five grade groups, 1 to 5. Grade group 1 (Gleason score ≤ 6) represents low or very low risk; grade groups 2 and 3 (Gleason score 3+4=7 and 4+3=7, respectively) represent intermediate risk; and grade groups 4 and 5 (Gleason score 8 and 9-10, respectively) represent high and very high risk. For each subject, the highest grade group detected by a given biopsy approach is assigned to that subject for that biopsy approach.
Time Frame: Up to 30 minutes
Population: Participants in whom cancer was detected by a given biopsy approach.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 13 | 22 | 23
units on a scale | 1.92 (1.04) | 1.86 (0.83) | 1.96 (1.15)
Statistical Analysis 1: Comparison: Acoustic Radiation Force Impulse (ARFI) vs MR-ultrasound Fusion vs Systematic Sampling; Test type: Other; p = 0.99, Kruskal-Wallis

4. Primary Outcome: Gleason Score
Description: A commonly used method to classify how cells appear in cancerous tissues; the less the cancerous cells look like normal cells, the more malignant the cancer; two numbers, each from 1 to 5, are assigned to the two most predominant types of cells present. These two numbers are added together to produce the Gleason score with a total range of 2 to 10. Higher numbers indicate more aggressive cancers. For each subject, the highest Gleason score detected by a given biopsy approach is assigned to that subject for that biopsy approach.
Time Frame: Up to 30 minutes
Population: Participants in whom cancer was detected by each biopsy approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 13 | 22 | 23
score on a scale | 6.62 (0.65) | 6.77 (0.61) | 6.74 (0.81)
Statistical Analysis 1: Comparison: Acoustic Radiation Force Impulse (ARFI) vs MR-ultrasound Fusion vs Systematic Sampling; Test type: Other; p = 0.74, Kruskal-Wallis

5. Primary Outcome: Number of Participants With Grade Group 1 Cancer, In Whom Cancer Was Detected
Description: The grading system has five grade groups, 1 to 5. Grade group 1 (Gleason score ≤ 6) represents low or very low risk; grade groups 2 and 3 (Gleason score 3+4=7 and 4+3=7, respectively) represent intermediate risk; and grade groups 4 and 5 (Gleason score 8 and 9-10, respectively) represent high and very high risk.
Time Frame: Up to 30 minutes
Population: Participants in whom Grade Group 1 was the highest grade of cancer that was detected by any biopsy approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 8 | 8 | 8
Participants | 2 | 6 | 6

6. Primary Outcome: Number of Participants With Grade Group 2 Cancer, In Whom Cancer (of Any Grade) Was Detected
Description: as for outcome 5
Time Frame: Up to 30 minutes
Population: Participants in whom Grade Group 2 was the highest grade of cancer that was detected by any biopsy approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 13 | 13 | 13
Participants | 7 | 12 | 11

7. Primary Outcome: Number of Participants With Grade Group 2 Cancer, Graded as Grade Group 2
Description: as for outcome 5
Time Frame: Up to 30 minutes
Population: Participants in whom Grade Group 2 was the highest grade of cancer that was detected by any biopsy approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 13 | 13 | 13
Participants | 3 | 11 | 8

8. Primary Outcome: Number of Participants With Grade Group 3 Cancer, In Whom Cancer (of Any Grade) Was Detected
Description: as for outcome 5
Time Frame: Up to 30 minutes
Population: Participants who were imaged with that biopsy approach and in whom Grade Group 3 was the highest grade of cancer that was detected by any biopsy approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 3 | 2 | 3
Participants | 1 | 1 | 3

9. Primary Outcome: Number of Participants With Grade Group 3 Cancer, Graded as Grade Group 3
Description: as for outcome 5
Time Frame: Up to 30 minutes
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 3 | 2 | 3
Participants | 1 | 0 | 2

10. Primary Outcome: Number of Participants With Grade Group 4 Cancer, In Whom Cancer (of Any Grade) Was Detected
Description: as for outcome 5
Time Frame: Up to 30 minutes
Population: Participants in whom Grade Group 4 was the highest grade of cancer that was detected by any biopsy approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 2 | 2 | 2
Participants | 2 | 2 | 2

11. Primary Outcome: Number of Participants With Grade Group 4 Cancer, Graded as Grade Group 4
Description: as for outcome 5
Time Frame: Up to 30 minutes
Population: Participants in whom Grade Group 4 was the highest grade of cancer that was detected by any biopsy approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 2 | 2 | 2
Participants | 0 | 1 | 2

12. Primary Outcome: Number of Participants With Grade Group 5 Cancer, In Whom Cancer (of Any Grade) Was Detected
Description: as for outcome 5
Time Frame: Up to 30 minutes
Population: Participants in whom Grade Group 5 was the highest grade of cancer that was detected by any biopsy approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 1 | 1 | 1
Participants | 1 | 1 | 1

13. Primary Outcome: Number of Participants With Grade Group 5 Cancer, Graded as Grade Group 5
Description: as for outcome 5
Time Frame: Up to 30 minutes
Population: Participants in whom Grade Group 5 was the highest grade of cancer that was detected by any biopsy approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
Number analyzed (Participants) | 1 | 1 | 1
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 30 mins
Description: Each participant was to undergo all three types of biopsy.
Groups:
- Systematic Sampling: Patients with suspected PCa who are scheduled to undergo an ultrasound fusion-MR prostate biopsy.
  Systematic sampling is a probability sampling method in which a random sample, with a fixed periodic interval, is selected from a larger population.
Arm/Group | Acoustic Radiation Force Impulse (ARFI) | MR-ultrasound Fusion | Systematic Sampling
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT04607135/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT04607135/ICF_000.pdf